CLINICAL TRIAL: NCT02317003
Title: Physical Exercise Prescription With PEdometeR in General Practice for Patients With Cardiovascular Risk Factors - The PEPPER Pragmatic Randomised Controlled Trial
Brief Title: Physical Exercise Prescription With PEdometeR in General Practice for Patients With Cardiovascular Risk Factors - PEPPER
Acronym: PEPPER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CHU-P 2014-04
Record Dates: First submitted 2014-12-10; First posted 2014-12-15 (Estimated); Last update posted 2022-08-02 (Actual); Status verified 2018-08

CONDITIONS: Sedentary Lifestyle; Cardiovascular Diseases; Hypertension; Hypercholesterolemia; Diabetes Mellitus, Type 2
Keywords: physical exercise; sedentarity; general practice; family medicine; pedometer
MeSH Terms: conditions — Sedentary Behavior; Cardiovascular Diseases; Hypertension; Hypercholesterolemia; Diabetes Mellitus, Type 2; Motor Activity | interventions — Prescriptions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention PPIL (Experimental): Intervention delivered by the family doctor and based on structured information delivery according to cognitive and behavioural theories, a personalised written physical activity prescription in number of steps per day, a pedometer, and a pedometer logbook similar to diabetes logbooks.
  Interventions: Behavioral: Intervention PPIL
- Control OR (Active Comparator): Oral recommendation of physical exercise delivered by the family doctor.
  Interventions: Behavioral: Control OR

INTERVENTIONS:
Behavioral: Intervention PPIL
  Other Names: Prescription, Pedometer, Information, Logbook
  Arms: Intervention PPIL
Behavioral: Control OR
  Other Names: Oral recommendation of physical exercise
  Arms: Control OR

SUMMARY:
This study evaluates the efficacy, in terms of energy expenditure, physical activity level, quality of life, blood pressure, waist circumference and weight, of a general practice based intervention involving a personalised physical exercise medical prescription, the structured delivery of information on the benefits of physical activity, a pedometer, and a pedometer log book, in 35 to 74 year old patients with cardiovascular risks factors.

DETAILED DESCRIPTION:
Background: Health benefits of physical activity have been shown to be at least as important as drug therapies in the prevention of cardiovascular diseases in patients with hypertension, hyperlipidaemia or diabetes. However, few strategies have demonstrated efficacy and practicality in the promotion of physical exercise among these high risk patients in general practice.

The PEPPER clinical study is a pragmatic randomised trial over a period of 12 months to evaluate the efficacy, in terms of physical activity level, of an intervention based on structured information delivery according to cognitive and behavioural theories, a personalised written physical activity prescription in number of steps per day, a pedometer, and a pedometer logbook similar to diabetes logbooks, in 35 to 74 year old patients with cardiovascular risks factors. This strategy will be compared to the commonly used oral recommendation of physical activity. The primary outcome is the change in total energy expenditure measured by accelerometry over a 7-day period. Secondary outcomes include changes in physical activity levels (International Physical Activity Questionnaire), quality of life (SF-36), blood pressure, weight, waist circumference, perceived obstacles to physical activity, and patient and doctors compliance with the suggested strategy. 140 patients will be recruited and followed up in 15 GP practices. Measures will be assessed at baseline, at 3 months and at 12 months (end of intervention).

The results of the PEPPER study are expected at the end of 2016. If the intervention proves effective in increasing durably the level of physical activity, this relatively simple and cheap strategy could help decrease the occurrence of cardiovascular events in a large high-risk population seen in general practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients consulting their general practitioner for a non-urgent matter
* with regular follow-up every 3 months for hypertension, hypercholesterolaemia or non insulin dependent type 2 diabetes.
* judged insufficiently active by their general practitioner based on negative answers to the questions : "Do you practice a physical activity or cycling more than an hour per week?" and "Does your occupation involve physical exertion?"

Exclusion Criteria:

* contraindication to moderate physical activity,
* non autonomous for walking,
* with cognitive or psychiatric impairment limiting the full understanding of the study,
* suffering from another limiting disease (coronary insufficiency, chronic cardiac failure, etc),
* who don't speak French,
* refusing to participate.

Ages: 35 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2015-03-16 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Change in total energy expenditure by accelerometry at 3 months compared to baseline | baseline and 12 weeks
  The total energy expenditure is measured with a wGT3x-BT Actigraph accelerometer worn at the belt during 7 consecutive days from morning to evening. It is measured in Metabolic Equivalent Task-Minutes per Week.

SECONDARY OUTCOMES:
Change in total energy expenditure by accelerometry at 12 months compared to baseline | baseline and 52 weeks
  The total energy expenditure is measured with a wGT3x-BT Actigraph accelerometer worn at the belt during 7 consecutive days from morning to evening. It is measured in Metabolic Equivalent Task-Minutes per Week.
Change in total energy expenditure by questionnaire at 3 months compared to baseline | baseline and 12 weeks
  The total energy expenditure is calculated with the self-administered International Physical Activity Questionaire (IPAQ) short version covering the past 7 days. It is expressed in Metabolic Equivalent Task-Minutes per Week.
Change in total energy expenditure by questionnaire at 12 months compared to baseline | baseline and 52 weeks
  The total energy expenditure is calculated with the self-administered International Physical Activity Questionaire (IPAQ) short version covering the past 7 days. It is expressed in Metabolic Equivalent Task-Minutes per Week.
Change in quality of life at 3 months compared to baseline | baseline and 12 weeks
  Change in quality of life as measured by the self-administered Short Form 36 questionnaire
Change in quality of life at 12 months compared to baseline | baseline and 52 weeks
  Change in quality of life as measured by the self-administered Short Form 36 questionnaire
Change in waist circumference at 3 months compared to baseline | baseline and 12 weeks
Change in waist circumference at 12 months compared to baseline | baseline and 52 weeks
Change in weight at 3 months compared to baseline | baseline and 12 weeks
Change in weight at 12 months compared to baseline | baseline and 52 weeks
Change in arterial blood pressure at 3 months compared to baseline | baseline and 12 weeks
Change in arterial blood pressure at 12 months compared to baseline | baseline and 52 weeks
Perceived obstacles to physical exercise | 52 weeks
  Perceived obstacles to physical exercise as measured by the Determinant of Physical Activity Questionnaire (DPAQ)
Adherence of doctors and patients to the suggested strategy | 12 weeks
Adherence of doctors and patients to the suggested strategy | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Denise Jolivot, MD, Study Chair — University Hospital, Angers; Laurent Connan, MD, Principal Investigator — Medical School, Angers
Locations (1):
- Angers University Hospital, Angers, France

REFERENCES:
- [Derived] Bellanger W, Peurois M, Connan L, Navasiolava N, Missud D, Py T, Begue C. Comparing physical activity prescription with verbal advice for general practice patients with cardiovascular risk factors: results from the PEPPER randomised controlled trial. BMC Public Health. 2023 Jul 20;23(1):1402. doi: 10.1186/s12889-023-16302-6. PMID 37475036
- [Derived] Missud DC, Parot-Schinkel E, Connan L, Vielle B, Huez JF. Physical activity prescription for general practice patients with cardiovascular risk factors-the PEPPER randomised controlled trial protocol. BMC Public Health. 2019 Jun 3;19(1):688. doi: 10.1186/s12889-019-7048-y. PMID 31159805